CLINICAL TRIAL: NCT07148089
Title: A Phase 1b, Multicenter, Open-Label, Dose Finding Study to Investigate the Safety and Tolerability of a Single Intravenous Dose of SGT-501 in Patients With Catecholaminergic Polymorphic Ventricular Tachycardia
Brief Title: A Study of SGT-501 Gene Therapy in Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT)
Acronym: ARTEMIS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Solid Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGT-501-101
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Catecholaminergic Polymorphic Ventricular Tachycardia
Keywords: Catecholaminergic polymorphic ventricular tachycardia (CPVT); SGT-501; Ryanodine Receptor 2 (RYR2); adeno-associated virus serotype 8 (AAV8); Cardiac; Gene Therapy
MeSH Terms: conditions — Polymorphic Catecholaminergic Ventricular Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (≥ 18 years of age) (Experimental): Participants will receive a single intravenous (IV) infusion (dose 1) of SGT-501.
  Interventions: Drug: SGT-501
- Cohort 2 (≥ 18 years of age) (Experimental): Participants will receive a single IV infusion (dose 2) of SGT-501.
  Interventions: Drug: SGT-501
- Cohort 3 (≥ 7 to < 18 years) (Experimental): Participants will receive a single IV infusion (level at or below dose(s) assessed in adults) of SGT-501.
  Interventions: Drug: SGT-501

INTERVENTIONS:
Drug: SGT-501 — IV for infusion

SUMMARY:
This is a Phase 1b, Multicenter, Open-Label, Dose Finding Study to Investigate the Safety and Tolerability of a Single Intravenous Dose of SGT-501 in participants with catecholaminergic polymorphic ventricular tachycardia (CPVT). The first-in-human (FIH) safety study will focus on obtaining safety data in adult participants. Cohort 1 and Cohort 2 (optional for dose exploration) will include participants ≥ 18 years of age. Cohort 3 will include participants ≥ 7 to < 18 years of age and will be initiated following data and safety monitoring board (DSMB) recommendations. Participants will be monitored for 5 years post-administration of SGT-501 including the active treatment period (1 year) and long-term follow-up (LTFU) (4 years) period.

ELIGIBILITY:
Inclusion Criteria:

Type of Participant and Disease Characteristics:

* Clinical diagnosis of CPVT, based on documented history of polymorphic or bidirectional non-sustained ventricular tachycardia with exercise or ventricular ectopy in a pattern consistent with CPVT on EST.
* Central Screening laboratory determination of a RYR2 variant that is pathogenic or likely pathogenic for CPVT.
* Documented history of life-threatening ventricular arrhythmic event defined as: survived sudden cardiac arrest, sudden cardiac arrest with appropriate implantable cardioverter defibrillator (ICD) shock, arrhythmic syncope, or sustained ventricular tachycardia (30 seconds or more) with or without ICD shock.
* On stable dose (defined as no change in dose by more than 50% for at least 1 month prior to Screening) of standard-of-care therapy defined as a beta-blocker and/or flecainide.
* Documented prior history of EST demonstrating a ventricular arrythmia score (VAS) score of ≥ 2.
* For the first 2 participants in each cohort only: a properly functioning ICD device in place. Following review of data from Cohorts 1 and 2, the Data Safety and Monitoring Board (DSMB) will determine if this criterion is required for participants in Cohort 3.
* Must be up to date with meningococcal vaccination per national guidelines or willing to receive meningococcal vaccine to achieve this.
* Other inclusion criteria to be applied as per protocol.

Exclusion Criteria:

* Abnormal liver function: gamma-glutamyl transferase (GGT) > 1.5 × upper limit of normal [ULN] or total bilirubin > ULN).
* Abnormal renal function defined by estimated glomerular filtration rate < 60 milliliter /minute (mL/min)/1.73-square meter (m^2) using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Formula.
* Clinically significant abnormalities of coagulation including international normalized ratio or activated partial thromboplastin time > 1.2 × ULN or platelets < 150,000 cells/cubic millimeter (mm^3).
* Potential concomitant cardiomyopathy or inherited arrhythmia as evidenced by pathogenic or likely pathogenic mutation other than RYR2 obtained on cardiac panel during Screening.
* Current or prior treatment with an approved or investigational gene transfer drug.
* Exposure to another investigational drug within 90 days prior to Screening or 5 half-lives since last administration, whichever is longer.
* Contraindication or unwillingness to receive required immunosuppression regimen.
* Body mass index ≥ 30 kilograms per square meter (kg/m^2).
* Other exclusion criteria to be applied as per protocol.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Event (TEAEs)s through Day 360 | First dose through Day 360

SECONDARY OUTCOMES:
Change from baseline in ventricular arrhythmia score (VAS) on exercise stress test (EST) at Day 180 | Baseline, Day 180
  An EST will be used to evaluate ventricular arrhythmia scores. The EST will be performed using the standard Bruce treadmill protocol.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No